CLINICAL TRIAL: NCT03722329
Title: A Randomised, Double-blind, Three-arm, Parallel Group, Single-dose Study to Compare the Pharmacokinetics, Safety, Tolerability, Immunogenicity, and Pharmacodynamics of Eculizumab (SB12, EU Sourced Soliris®, and US Sourced Soliris®) in Healthy Subjects
Brief Title: Pharmacokinetic, Safety, Tolerability, Immunogenicity, and Pharmacodynamic Study of SB12 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SB12-1001
Record Dates: First submitted 2018-10-24; First posted 2018-10-26 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Healthy
MeSH Terms: interventions — eculizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- SB12 (Experimental): SB12 (proposed eculizumab biosimilar)
  Interventions: Drug: Eculizumab
- EU Soliris (Active Comparator): EU sourced Soliris (eculizumab)
  Interventions: Drug: Eculizumab
- US Soliris (Active Comparator): US sourced Soliris (eculizumab)
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — Eculizumab Injection. 300 mg, single dose

SUMMARY:
This study is to evaluate PK, safety, tolerability, immunogenicity, and PD profiles of SB12, EU sourced Soliris, and US sourced Soliris in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Have a body weight between 70-95 kg and a body mass index between 20.0-29.9 kg/m²
* Have systolic blood pressure (SBP) ≤ 140 and ≥ 90 mmHg, diastolic blood pressure (DBP) ≤ 95 and ≥ 45 mmHg, and pulse rate ≥ 40 and ≤ 100 beats per minute or assessed as not clinically significant
* Have physical examination and 12-lead ECG results without clinically significant finding at Screening and Day -1 visits
* Non-smoker or smoker whose daily smoking does not exceed 10 cigarettes, 3 cigars, or 3 pipes for at least 30 days prior to Screening visit. Subjects should agree to abstain from smoking while resident at the clinical study site.
* Willing to receive vaccination against N. meningitidis at least 14 days prior to IP administration
* Male subjects must be willing to abstain from sexual intercourse or willing to use a condom in addition to having their female partner use another form of contraception unless their partner is infertile from the time of IP administration until 5 months after IP administration
* Must be willing and able to comply with scheduled visits, treatment plan, clinical laboratory tests, and other study procedures including lifestyle considerations
* Have competence in speaking, writing and comprehending the local language where the study is conducted

Exclusion Criteria:

* Have a history/presence of clinically significant atopic allergy, allergic/hypersensitive reactions, or known or suspected clinically relevant drug hypersensitivity to eculizumab or its excipients
* Contraindication for IP or non-IP to be used in the study
* History of N. meningitidis infection
* Known or suspected hereditary or acquired complement deficiency
* Clinically significant active infection within 28 days before IP administration
* Any systemic or local infection, a known risk for developing sepsis and/or known active inflammatory condition
* Have previously been exposed to eculizumab (Soliris and its biosimilar)
* Previous treatment with a monoclonal antibody or fusion protein within 9 months prior to IP administration and/or have an evidence of immunogenicity from previous exposure to a monoclonal antibody or fusion protein
* Have previously been exposed to an immunosuppressive agent or biological agent (any other than a monoclonal antibody or fusion protein) within 120 days prior to IP administration
* Any of the following abnormal laboratory values at Screening and Day -1 visits:

  1. Serum alanine transaminase and/or aspartate transaminase ≥ 1.5 × ULN
  2. Serum C-reactive protein ≥ 10 mg/L
  3. Serum creatinine > 1.5 × ULN
  4. Whole blood cell count < 3000/mm3, absolute lymphocyte count < 800/mm3, and/or absolute neutrophil count ≤ 1500/mm3
  5. Any other laboratory abnormalities assessed as clinically significant by the Investigator
* Positive test result for hepatitis B surface antigen and/or hepatitis B core antibody, hepatitis C virus antibody, or human immunodeficiency virus at Screening
* Surgery within 90 days prior to IP administration, and/or operation during study period
* Average intake of alcoholic beverages of more than 21 units/week for males and 14 units/week for females
* Drug abuse or a positive urinary drug screening result
* Have any prescription medicine or over-the-counter medicines (except paracetamol) that might have an effect on the objectives of the study, within 14 days prior to IP administration
* Donated >100 mL blood or plasma within 28 days prior to IP administration
* Subject directly involved in the conduct of the clinical study
* Vulnerable subjects
* Pregnant or nursing (lactating) women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
AUCinf | Day 1 to Day 64
  Area under the concentration-time curve from time zero to infinity

SECONDARY OUTCOMES:
AUClast | Day 1 to Day 64
  Area under the concentration-time curve from time zero to the last quantifiable concentration
Cmax | Day 1 to Day 64
  Maximum observed serum concentration
Tmax | Day 1 to Day 64
  Time to reach Cmax
Vz | Day 1 to Day 64
  Volume of distribution during terminal phase
λz | Day 1 to Day 64
  Terminal rate constant
T1/2 | Day 1 to Day 64
  Terminal half-life
Clearance | Day 1 to Day 64
  Total body clearance
%AUCextrap | Day 1 to Day 64
  Percentage of AUCinf due to extrapolation from time of last measurable concentration (Tlast) to infinity
Incidence of Treatment-Emergent Adverse Events | Day 1 to Day 64
  Experience at least 1 treatment-emergent adverse event
Incidence of Serious Adverse Events | Day 1 to Day 64
  Experience at least 1 serious adverse event
Incidence of ADA | Day 1 to Day 64
  Incidence of anti-drug antibodies
Incidence NAb | Day 1 to Day 64
  Incidence neutralising antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Rainard Fuhr, MD, Principal Investigator — PAREXEL International GmbH, Early Phase Clinical Unit - Berlin
Locations (1):
- PAREXEL International GmbH, Early Phase Clinical Unit - Berlin, Berlin, Germany